CLINICAL TRIAL: NCT03459534
Title: A Phase 3 Multinational, Multi-center, Single-arm, Open-label Study for the Efficacy and Safety of Radotinib in Ph+ Chronic Phase Chronic Myeloid Leukemia Patients With Failure or Intolerance to Previous TKIs Therapy Including Imatinib
Brief Title: A Phase 3 Study for the Efficacy and Safety of Radotinib in CP-CML Patients With Failure or Intolerance to Previous TKIs
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT51KRI03; 2018-003810-42 (EudraCT Number)
Record Dates: First submitted 2018-02-12; First posted 2018-03-09 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2023-10

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase; CML, Chronic Phase; CML, Refractory; CML - Philadelphia Chromosome
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radotinib HCl (Experimental): Enrolled subjects will continue to administer Radotinib 400mg twice daily (800mg/day) orally every 12 hours at regular dosing hours for 12 months.
  Dose modification is allowed if the subject cannot comply with the protocol-defined dosing schedule due to hematologic or non-hematologic toxicities and toxicities resolve within 28 days (within 42 days for hematologic toxicities). For radotinib, maximum 2 dose reductions will be allowed by stage to 600mg and to 400mg.
  Interventions: Drug: Radotinib HCl

INTERVENTIONS:
Drug: Radotinib HCl — 1. Brand name/manufacturer: Supect Cap./IL-YANG PHARM. Co., Ltd.
  2. Active ingredient: radotinib HCl 106.8mg (100mg as radotinib) or HCl 213.6mg (200mg as radotinib)
  3. Appearance and formulation: hard capsule with a light blue cap and a body containing pale yellow powder
  4. Storage conditions: Store in an airtight light proof container at room temperature.
  Other Names: SUPECT

SUMMARY:
In a multinational, multicenter, single-arm, open-label and Phase III Radotinib clinical study, chronic phase Ph+ chronic myeloid leukemia patients with failure or intolerance to previous TKIs therapy including Imatinib will be recruited. In this phase 3 study, 173 subjects are expected to be enrolled in a single arm with the administration of Radotinib 400mg twice daily, which includes 10% of dropout rate.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years old
2. Chronic Phase Ph+ Chronic Myeloid Leukemia patients who failed or intolerance the previous TKIs therapy including Imatinib Imatinib
3. ECOG scale 0, 1 or 2
4. Chronic phase is defined as all of the following conditions that subjects meet.

   * Blast in peripheral blood and bone marrow <15%
   * The sum of blast and promyelocyte in peripheral blood and bone marrow <30%
   * Basophil in peripheral blood <20%
   * Platelets count ≥50 × 10^9/L (≥ 50,000/mm3) (But, transient prior therapy related thrombocytopenia [< 50 × 109/L (< 50,000/mm3)] is acceptable
   * No evidence of involvement of extramedullary leukemia other than enlargements of liver and spleen
5. Patients who have adequate organ functions as defined below:

   * Total bilirubin < 1.5 × upper limit of normal (ULN)
   * SGOT and SGPT < 2.5× ULN
   * Creatinine < 1.5 × ULN
   * Serum amylase and lipase ≤ 1.5 × ULN
   * Alkaline Phosphatase ≤ 2.5 × ULN (only if not related to the tumor)
6. Women of childbearing potential should have a negative serum or urine pregnancy test within 14 days of the enrollment.
7. Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 1 month (4 weeks) after the last dose of investigational product in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

1. Patients who have been diagonised accelerated phase and blast crisis CML in previous therapy if only once.
2. Patients with CCyR at the time of screening
3. Any below impaired cardiac function:

   * LVEF <45% or < lower bound of normal limit of study site (whichever higher), confirmed by echocardiogram at the site
   * Patients who cannot have QT intervals measured according to ECG
   * Complete left bundle branch block
   * Patients with cardiac pacemakers
   * Patients with congenital long QT syndrome or the family history of known long QT syndrome
   * History of, or presence of symptomatic ventricular or atrial tachyarrhythmias
   * Clinically significant resting bradycardia (< 50 bpm)
   * The mean QTcF >450msec following three consecutive ECG tests at baseline

     : Screening test will be performed again for QTcF after the adjustment of electrolyte if QTcF >450msec and the electrolyte is not within the normal range.
   * Medical history of clinically confirmed myocardial infarction
   * Medical history of unstable angina (within last 12 months)
   * Other clinically significant cardiac disease
4. Patients with T315I point mutations
5. Patients with central nervous system involvement as cytopathologically confirmed
6. Severe or uncontrolled chronic disease
7. Significant medical history of congenital or acquired bleeding disorders that are not related to leukemia
8. Patients who previously received radiotherapy to at least 25% of the bodies with high portion of bone marrow
9. Patients who received the major surgery within 4 weeks before the initiation of the IP administration or who failed to recover from the surgery that was performed before then.
10. Patients who participated in other clinical study and are receiving any other IP.
11. Patients who cannot give consent to the clinical study.
12. Patients who have concurrently clinically significant primary malignancy
13. Patients currently receiving treatment with a strong CYP3A4 inhibitors or strong CYP3A4 inducers or therapeutic Cumarin derivatives and that can neither stop the administration of these drugs before the start of the IP administration nor switch to other drugs.
14. Patients who are currently receiving treatment with a medication that has the potential to prolong QT intervals and can neither stop the administration of the drugs before the start of the IP administration nor switch to other drugs. If subjects need to start such drug treatments during the study, they should contact the sponsor, IL-YANG PHARM. Co., Ltd.
15. Gastrointestinal disorder or gastrointestinal disease that may result in a significant change in the absorption of the investigational product
16. Medical history of acute or chronic pancreatitis within the past one year
17. Acute or chronic liver, pancreas, or severe kidney disease that are not associated with the disease
18. Patients known seropositive to human immunodeficiency virus (HIV), current acute or chronic hepatitis B (hepatitis B surface-antigen positive), hepatitis C, or cirrhosis. Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA < 500 IU/mL or site specific local lab normal range lower limit assessed by investigator), and cured hepatitis C patients can be enrolled.
19. Women patients that meet the following conditions should be excluded from the clinical study.

    * Pregnancy
    * Breastfeeding
    * Pregnancy confirmed at screening pregnancy test
    * Women of childbearing potential who is unwilling to use an appropriate method of contraception during the study
20. Men patients who are unwilling to use and appropriate method of contraception during the study
21. Patients who have hypersensitivity to active ingredient or any of the excipients of this investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Cytogenetic Response (MCyR) | at month 6
  MCyR is defined as 0~35% CCyR+PCyR based on ≥20 metaphase myelocytes. Chromosome test results from <20 metaphase myelocytes will be excluded from the analysis.

SECONDARY OUTCOMES:
Cytogenetic Response (CCyR) | at month 12/24, by month 24
  CCyR is defined as complete loss of Ph chromosome based on ≥20 metaphase myelocytes. Chromosome test results from <20 metaphase myelocytes will be excluded from the analysis.
Major molecular response | at month 12/24, by month 24
  MMR is defined as a ≥3-log reduction in BCR-ABL1 transcript level from the standardized reference or BCR-ABL1/ABL % of ≤0.1% according to the international reference when the level of BCR-ABL1 gene was measured by RQ-PCR, a standardized quantitative genetic method.
Overall Survival(OS) | by month 24
  OS is defined as the duration from the first day of Radotinib administration to the day of death for certain causes.
Progression Free Survival (PFS) | by month 24
  PFS is defined as the duration from the first day of Radotinib administration to the earliest day of disease progression or death for certain causes.

OTHER OUTCOMES:
BCR-ABL1 point mutation | up to month 24
  Incidence rate of BCR-ABL1 point mutations that are newly found during the course of radotinib treatment
correlation between the concentration of radotinib in blood and the response (efficacy and safety) | up to month 24
  To measure the concentration of radotinib in blood
Incidence of Radotinib-Adverse Events | up to month 24
  Toxicities will be evaluated in all subjects treated with radotinib.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wook Kim, Principal Investigator — the Catholic University of Korea's St. Mary's Hospital
Locations (17):
- Russia (5):
  - Territorial State Budgetary Institution, Barnaul
  - Federal State Budgetary Institution of Science, Kirov
  - Federal State Budgetary Institution, Moscow
  - Hematology Centre based on City Clin. Hosp. n.a. S.P. Botkin, Moscow
  - Federal State Budgetary Institution, Saint Petersburg
- Uijeongbu Eulji Medical Center, Eulji University, Uijeongbu-si, Gyeonggi-do, South Korea
- Turkey (Türkiye) (6):
  - Ankara University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Mersin University Medical Faculty, Mersin
  - Ondokuz Mayis Univ. Med. Fac., Samsun
- Ukraine (5):
  - CI Cherkasy Regional Oncological Dispensary of CRC, Cherkassy
  - CTPI Chernihiv Regional Oncological Dispensary, Chernihiv
  - CI Dnipropetrovsk CMCH #4 OF Dnipropetrovsk RC, Dnipro
  - Institute of CR of SI NSC of Radiation Medicine of NAMSU H&T Unit, Kyiv
  - SI Institute of Blood Pathology and Transfusion Medicine of AMSU, Lviv

IPD SHARING:
Plan to Share IPD: No